CLINICAL TRIAL: NCT02998619
Title: Retrospektive Analyse Der Radiotherapie Des Pelvinen Lymphabflusses Beim Lokalisierten Prostatakarzinom Vom Hochrisikotyp Anhand Der Klinikdatenbank 2010-2016
Brief Title: Radiotherapy of Pelvic Lymph Nodes in High Risk Prostate Cancer - A Retrospective Analysis
Status: Completed | Type: Observational
Sponsor: Kantonsspital Graubuenden (Other)
Responsible Party: Sponsor
Other Study IDs: BASEC 2016-01325
Record Dates: First submitted 2016-12-11; First posted 2016-12-20 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Prostatic Neoplasms Benign; Radiotherapy Side Effect; Lymph Node Disease
MeSH Terms: conditions — Radiation Injuries | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Radiotherapy: Radiation to prostate/seminal vesicles including pelvic lymph nodes Postoperative radiation to prostate bed including pelvic lymph nodes
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Radiation to prostate/seminal vesicles including pelvic lymph nodes Postoperative radiation to prostate bed including pelvic lymph nodes

SUMMARY:
Men with high risk prostate cancer who underwent radiotherapy of the prostate/seminal vesicles or underwent postoperative radiotherapy including pelvic lymph nodes between 2010 and 2016 are analyzed retrospectively. The aims are to estimate progression-free survival as well as toxicity according to CTCAE v4.03.

DETAILED DESCRIPTION:
Collection of data and retrospective analysis of patients with high risk prostate cancer treated with radiotherapy to pelvic lymph nodes.

What influence has irradiation of pelvic lymph nodes on patients with high risk prostate cancer in terms of progression free survival and toxicity. How does this influence side effects with respect to gastrointestinal (proctitis, abdominal pain, diarrhea) and genitourinary (cystitis, urinary disorders) toxicities (CTCAE v4.03)

ELIGIBILITY:
Inclusion Criteria:

* Men with high risk prostate cancer treated with radiotherapy to prostate/seminal vesicles or postoperative radiotherapy and pelvic lymph nodes at the Kantonssptial Graubuenden, Department of Radiation Oncology between 2010 and 2016

Exclusion Criteria:

* Men with prostate cancer other than high risk disease and no radiotherapy to pelvic lymph nodes

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective analysis of men irradiated for high risk prostate cancer including pelvic lymph nodes (L5/S1)
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2016-12; Primary Completion 2017-11-11 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | through study completion, an average of 2 years
  PSA progession-free survival will be measured

SECONDARY OUTCOMES:
Toxicity (CTCAE v4.03) | through study completion, an average of 2 years
  GI, GU Toxicities as well as Erectile Dysfunction will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Zwahlen, MD, MBA, Study Chair — Kantonsspital Graubuenden
Locations (1):
- Kantonsspital Graubuenden, Chur, Switzerland

IPD SHARING:
Plan to Share IPD: No